CLINICAL TRIAL: NCT00814385
Title: A Randomized, Partially Observer-blind, Single-centre Study to Evaluate Safety and Immunogenicity of MF59-adjuvanted or Non-adjuvanted H5N1 Influenza Vaccines in Adults Primed With Adjuvanted Influenza A/Vietnam/1194/04 (H5N1) Vaccine
Brief Title: Immunogenicity of Adjuvanted or Non-adjuvanted H5N1 Booster Vaccine in Adults Primed to A/VN/1194/04
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University Hospitals, Leicester (Other)
Collaborators: Medical Research Council (Other Government); Novartis (Industry); Public Health England (Other Government); National Institute of Biological Standards and Control (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double
Other Study IDs: UHL10492
Record Dates: First submitted 2008-12-23; First posted 2008-12-24 (Estimated); Last update posted 2014-06-03 (Estimated); Status verified 2014-06

CONDITIONS: Influenza
MeSH Terms: conditions — Influenza, Human | interventions — PRIME protocol

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (9):
- Vaccine arm 1 (Active Comparator): Mf59-adjuvanted A/VN/1194/04 H5N1 vaccine containing 7.5microg haemagglutinin, given as single dose followed by non-adjuvanted H5N1 clade 2 vaccine containing 3.75microg dose at 52 weeks
  Interventions: Biological: Aflunov (Single prime, single boost)
- Vaccine arm 2 (Active Comparator): Mf59-adjuvanted A/VN/1194/04 H5N1 vaccine containing 7.5microg haemagglutinin, given as single dose followed by MF59-adjuvanted H5N1 clade 2 vaccine containing 3.75microg dose at 52 weeks
  Interventions: Biological: Aflunov (Single prime, single boost)
- Vaccine arm 3 (Active Comparator): Mf59-adjuvanted A/VN/1194/04 H5N1 vaccine containing 7.5microg haemagglutinin, given as single dose followed by non-adjuvanted H5N1 clade 2 vaccine containing 7.5microg dose at 52 weeks
  Interventions: Biological: Aflunov (single prime, single boost)
- Vaccine arm 4 (Active Comparator): Mf59-adjuvanted A/VN/1194/04 H5N1 vaccine containing 7.5microg haemagglutinin, given as single dose followed by MF59-adjuvanted H5N1 clade 2 vaccine containing 7.5microg dose at 52 weeks
  Interventions: Biological: Aflunov (single prime, single boost)
- Vaccine arm 5 (Active Comparator): Two doses of Mf59-adjuvanted A/VN/1194/04 H5N1 vaccine containing 7.5microg haemagglutinin followed by non-adjuvanted H5N1 clade 2 vaccine containing 3.75microg dose at 52 weeks
  Interventions: Biological: Aflunov (Double prime, single boost)
- vaccine arm 6 (Active Comparator): Two doses of Mf59-adjuvanted A/VN/1194/04 H5N1 vaccine containing 7.5microg haemagglutinin followed by MF59-adjuvanted H5N1 clade 2 vaccine containing 3.75microg dose at 52 weeks
  Interventions: Biological: Aflunov (double prime, single boost)
- Vaccine arm 7 (Active Comparator): Two doses of Mf59-adjuvanted A/VN/1194/04 H5N1 vaccine containing 7.5microg haemagglutinin followed by non-adjuvanted H5N1 clade 2 vaccine containing 7.5microg dose at 52 weeks
  Interventions: Biological: Aflunov (double prime, single boost)
- Vaccine arm 8 (Active Comparator): Two doses of Mf59-adjuvanted A/VN/1194/04 H5N1 vaccine containing 7.5microg haemagglutinin followed by MF59-adjuvanted H5N1 clade 2 vaccine containing 7.5microg dose at 52 weeks
  Interventions: Biological: Aflunov (double prime, single boost)
- Vaccine arm 9 (Active Comparator): No priming dose and single dose MF59 adjuvanted H5N1 vaccine at 52 weeks
  Interventions: Biological: Aflunov (No prime, single boost)

INTERVENTIONS:
Biological: Aflunov (Single prime, single boost) — Priming with single dose 7.5microg MF59-adjuvanted A/VN/1194/04 then non-adjuvanted H5N1 vaccine containing 3.75microg at 52 weeks
  Other Names: Aflunov
  Arms: Vaccine arm 1
Biological: Aflunov (Single prime, single boost) — Priming with single dose 7.5microg MF59-adjuvanted A/VN/1194/04 then MF59-adjuvanted H5N1 vaccine containing 3.75microg at 52 weeks
  Other Names: Aflunov
  Arms: Vaccine arm 2
Biological: Aflunov (single prime, single boost) — Priming with single dose 7.5microg MF59-adjuvanted A/VN/1194/04 then non-adjuvanted H5N1 vaccine containing 7.5microg at 52 weeks
  Other Names: Aflunov
  Arms: Vaccine arm 3
Biological: Aflunov (single prime, single boost) — Priming with single dose 7.5microg MF59-adjuvanted A/VN/1194/04 then MF59-adjuvanted H5N1 vaccine containing 7.5microg at 52 weeks
  Other Names: aflunov
  Arms: Vaccine arm 4
Biological: Aflunov (Double prime, single boost) — Priming with two doses 7.5microg MF59-adjuvanted A/VN/1194/04 then non-adjuvanted H5N1 vaccine containing 3.75microg at 52 weeks
  Other Names: aflunov
  Arms: Vaccine arm 5
Biological: Aflunov (double prime, single boost) — Priming with two doses 7.5microg MF59-adjuvanted A/VN/1194/04 then MF59-adjuvanted H5N1 vaccine containing 3.75microg at 52 weeks
  Other Names: aflunov
  Arms: vaccine arm 6
Biological: Aflunov (double prime, single boost) — Priming with two doses 7.5microg MF59-adjuvanted A/VN/1194/04 then non-adjuvanted H5N1 vaccine containing 7.5microg at 52 weeks
  Other Names: aflunov
  Arms: Vaccine arm 7
Biological: Aflunov (double prime, single boost) — Priming with two doses 7.5microg MF59-adjuvanted A/VN/1194/04 then MF59-adjuvanted H5N1 vaccine containing 7.5microg at 52 weeks
  Other Names: aflunov
  Arms: Vaccine arm 8
Biological: Aflunov (No prime, single boost) — No Priming then MF59-adjuvanted H5N1 vaccine containing 7.5microg at 52 weeks
  Other Names: aflunov
  Arms: Vaccine arm 9

SUMMARY:
This study focuses on pre-pandemic priming of man against H5 influenza with the goal of mounting a robust antibody response to small quantities of vaccine either before or during an H5 pandemic.

DETAILED DESCRIPTION:
OBJECTIVES:

Immunogenicity objectives

1. To evaluate the magnitude of the antibody responses to one or two 'priming' 0.5mL intramuscular (IM) doses of an MF59-adjuvanted A/Vietnam/1194/2004 (H5N1 Clade 1) influenza vaccine, each dose containing 7.5μg of H5N1 haemagglutinin, in immunologically naïve subjects;
2. To examine the kinetics of the antibody responses to one 0.5mL 'booster' intramuscular dose of antigenically drifted MF59-adjuvanted vaccine, or non-adjuvanted antigenically drifted vaccine, given at doses of 3.75 or 7.5μg, in subjects primed with one or two doses of an MF59-adjuvanted A/Vietnam/1194/2004 (H5N1 Clade 1) influenza vaccine;
3. To evaluate the magnitude of the antibody responses to one 0.5mL 'booster' intramuscular dose of antigenically drifted MF59-adjuvanted vaccine, or non-adjuvanted antigenically drifted vaccine, given at doses of 3.75μg or 7.5μg, in subjects primed with one or two doses of an MF59-adjuvanted A/Vietnam/1194/2004 (H5N1 Clade 1) influenza vaccine;
4. To evaluate the breadth of the antibody responses induced by 'priming' (see 1., above), and 'booster' vaccination regimens (see 2., and 3., above), with respect to a representative range of antigenically distinct H5N1 viruses (wild-type and attenuated); and
5. To evaluate the persistence of the antibody responses induced by 'priming' (see 1., above), and 'booster' vaccination regimens (see 2., and 3., above).

Safety objective

1. To evaluate the safety of the administration of one or two 'priming' 0.5mL intramuscular (IM) doses of an MF59-adjuvanted A/Vietnam/1194/2004 (H5N1 Clade 1) influenza vaccine (each dose containing 7.5μg of H5N1 haemagglutinin), in immunologically naïve subjects, followed by one 3.75μg or 7.5μg 'booster' dose of antigenically drifted MF59-adjuvanted H5N1 vaccine, or non-adjuvanted antigenically drifted H5N1 vaccine.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects 18 to 59 years of age, or 60 years of age and older, mentally competent, who have signed an informed consent form after having received a detailed explanation of the study protocol;
2. Are in good health or have one or more stable (See footnote) medical conditions, as determined by:

   1. Medical history,
   2. Physical examination,
   3. Clinical judgment of the medical investigator;
3. Are able to understand and comply with all study procedures and to complete study diaries, can be contacted, and will be available for study visits.
4. Subjects who experienced fever (defined as axillary temperature >38oC) within 3 days prior to Visit 1;
5. Subjects who are pregnant or breastfeeding;
6. Females of childbearing potential who refuse to use an acceptable method of birth control for a period of 56 days before and after each vaccination. Adequate contraception is defined as hormonal (e.g., oral, injection, transdermal patch, implant, cervical ring), barrier (e.g., condom with spermicide or diaphragm with spermicide), intrauterine device (e.g., IUD), monogamous relationship with vasectomised partner who has been vasectomised for 6 months or more prior to the subject's study entry, or abstain from heterosexual intercourse (e.g., through sexual orientation or religious or other beliefs about premarital intercourse);
7. Subjects with any serious disease, including:

   1. cancer,
   2. acute or progressive hepatic disease,
   3. acute or progressive renal disease,
   4. chronic pulmonary disease requiring home oxygen therapy,
   5. active neurological disorder,
   6. autoimmune disease (including rheumatoid arthritis);
8. Subjects for whom surgery is planned during the study period;
9. Subjects with a bleeding diathesis;
10. Subjects with hypersensitivity to eggs, chicken protein, chicken feathers, influenza viral protein, neomycin or kanamycin, or any other component of the study vaccine;
11. Subjects with a history of any neurological symptoms and signs, or anaphylactic shock following administration of any vaccine;
12. Subjects with known or suspected impairment/alteration of immune function, for example, resulting from:

    1. receipt of oral immunosuppressive therapy (e.g., corticosteroid therapy or cancer chemotherapy) (long-term, inhaled steroids for asthma management is acceptable),
    2. receipt of immunostimulants or interferon,
    3. receipt of parenteral immunoglobulin preparation, blood products, and/or plasma derivatives within 3 months prior to Visits 1 (Day 1), 2 (Day 22), or 5 (Day 382), or planned during the full length of the study,
    4. high risk from developing an immunocompromising disease;
13. Actual or planned receipt of another vaccine during the period 3 weeks before to 3 weeks after vaccination on Days 1, 22, and 382;
14. Subjects with a history of (or current) drug or alcohol abuse (20g/day for females; 30g/day for males) that in the investigator's opinion would interfere with safety of the subject or the evaluation of the study objectives;
15. Subjects who are unable to lead an independent life either physically or mentally;
16. Have participated in a previous study of H5 avian influenza vaccine;
17. Have been previously vaccinated with a vaccine containing MF59 or similar adjuvant;
18. Subjects with any condition, which, in the opinion of the Investigator, might interfere with the evaluation of the study objectives.

Exclusion Criteria:

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 606 (Actual)
Dates: Start 2008-11; Primary Completion 2013-09 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Geometric mean antibody titres to influenza H5N1 by neutralising antibody, HI and SRH | pre vaccination, 3 weeks, 6 weeks, 52 weeks, 55 weeks, 56 weeks

SECONDARY OUTCOMES:
local and systemic reactogenicity | within 7 days of each vaccination
Seroprotective and seroconversion responses to H5N1 by neutralising antibody, HI and SRH | Prevaccination, 3 weeks, 6 weeks, 52 weeks, 55 weeks and 56 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Karl G Nicholson, FRCP, MD, Principal Investigator — University of Leicester
Locations (2):
- United Kingdom (2):
  - University Hospitals Leicester, Leicester, Leicestershire
  - Clincal Trials Unit Leicester Royal Infirmary, Leicester